CLINICAL TRIAL: NCT04566432
Title: Therapeutic ResistAnce and Clonal Evolution Assessed With Liquid Biopsy of NSCLC Patients Treated With Immune Checkpoint Inhibitors (ICIs) or Targeted Therapy
Brief Title: Therapeutic ResistAnce and Clonal Evolution Assessed With Liquid Biopsy in ICIs Treated NSCLC Patients
Status: Recruiting | Type: Observational
Sponsor: Geneplus-Beijing Co. Ltd. (Industry)
Collaborators: Shanghai Chest Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TRACELib002
Record Dates: First submitted 2020-07-23; First posted 2020-09-28 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Lung Neoplasms; Lung Cancer, Nonsmall Cell; Adenocarcinoma of Lung; Squamous Cell Lung Cancer
Keywords: Next Generation Sequencing (NGS); Liquid biopsy; Immune Checkpoint Inhibitor; Whole Transcriptome Sequencing
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood (including plasma, white cells), tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immune checkpoint inhibitors
  Interventions: Other: Observation
- Targeted therapy: Targeting ALK, ROS1, MET ex14 skipping
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — observe the association of ctDNA with efficacy of treatment

SUMMARY:
To evaluate the predictive value of ctDNA in response, relapse for patients treated with immune checkpoint inhibitors or targeted therapy for ALK, ROS1, MET ex14 skipping.

DETAILED DESCRIPTION:
In the study, 250 advanced NSCLC patients will be recruited. All the patients will receive tissue biopsy and circultating tumor DNA (ctDNA) liquid biopsy before entry the study. Patients who have no actionable mutations in EGFR or ALK and receive ICIs treatment and patients who carry actionable ROS1 fusion, ALK fusion or MET exon 14 skipping mutation and receive TKI treatment according to guidelines will take liquid biopsy assay to monitor the mutation status. The study will be ended when over 70% of the patients had a progressive disease (PD) in their targeted lesion.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Newly diagnosed and histological or cytological confirmed stage IIIB-IV lung adenocarcinoma or squamous cell carcinoma patients according to the AJCC staging system. The stage IV lung cancer and brain metastasis can be diagnosed by imaging and enhanced CT respectively
* No EGFR mutation in tissue and ctDNA
* Received immune checkpoint inhibitors as the first line therapy
* ECOG performance status 0-2 with expected more than 6 months of survival time
* Willingness to comply with required protocols and give permission to use the data for clinical research and products development

Exclusion Criteria:

* Patients have other primary cancers
* Patients have symptomatic brain metastasis, complications that are associated with brain metastasis or cognitive disorders
* Patients failed in either plasma or tissue sample QC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: treatment naïve Stage IIIB or Stage IV NSCLC patients, adenocarcinoma or squamous cell carcinoma
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
the evolution of ctDNA mutation profile during treatment | every 2-3 cycles of treatment upon physicians' request, ctDNA mutation analysis and clonal analysis (each cycle is 28 days)
  ctDNA mutation will be detected, PyClone based clonal analysis will be performed to analyze the clonal dominance

SECONDARY OUTCOMES:
Resistant mechanisms of targeted therapy | At the time of disease progression (through study completion, an average of 1.5 years)
  Resistant mutations will be identified from ctDNA or tissue mutations

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided